CLINICAL TRIAL: NCT06766851
Title: Comparison of Single-Needle Arthrocentesis and Intravenous Catheter-Assisted Arthrocentesis in the Management of Temporomandibular Joint Disorders
Brief Title: Evaluation of the Effectiveness of Arthrocentesis Using Catheter in the Treatment of Temporamandibular Joint Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Gorkem Tekin, Asst.Prof., Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EskisehirOU-TEKIN-002
Record Dates: First submitted 2025-01-04; First posted 2025-01-09 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: TMJ Disc Disorder; Treatment; Arthrocentesis
Keywords: Branul

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Catheter group (Experimental): Patients presenting temporomandibular joint disc displacement without reduction (DDwoR) treated with catheter arthrocentesis. The upper joint space was entered with a 16 gauge 45 mm long branul. The 16 gauge metal cannula was removed and the plastic sheath was left in the upper joint space. The 18 gauge metal cannula, which was 1 size smaller, was placed inside the sheath. The irrigation solution was administered through the 18 gauge metal cannula and the irrigation solution flowed out of the space between the cannula and the sheath + I-PRF
  Interventions: Other: Procedure: TMJ Arthrocentesis
- conventional single needle group (Active Comparator): Patients presenting temporomandibular joint disc displacement without reduction (DDwoR) treated with single puncture arthrocentesis + I-PRF
  Interventions: Other: Procedure: TMJ Arthrocentesis

INTERVENTIONS:
Other: Procedure: TMJ Arthrocentesis — Temporomandibular joint arthrocentesis

SUMMARY:
The study focused on arthrocentesis performed using a catheter, aiming to assess its effects on pain perception and mouth opening in patients with TMJ disorders.

DETAILED DESCRIPTION:
Two groups will be formed consisting of patients who present with complaints of TMJ pain, limited mouth opening and hearing sounds in the joint and are diagnosed with TMJ disorder. After explaining the I-PRF protocol obtained by taking blood to both groups and obtaining the necessary consents, arthrocentesis will be performed on the relevant joint area using a catheter for the patients in the first group and a single needle for the patients in the second group. Patients will be called for check-ups on the 1st day, 1st week and 1st month after the protocols and the current perceived pain level before and after the treatment will be determined by scoring with Visual Analog Scala (VAS) and measuring the mouth opening with a ruler ( mm).

ELIGIBILITY:
Patients included in this study were adult individuals aged 18 years and older who were diagnosed with stage 3 or higher temporomandibular joint (TMJ) disorder according to the Wilkes classification, based on magnetic resonance imaging (MRI) in addition to clinical evaluation. Eligible patients had unilateral internal TMJ disorder and exhibited clinical symptoms such as TMJ-related pain and/or joint sounds, and limited mouth opening. Furthermore, only patients whose symptoms persisted despite at least one month of occlusal splint therapy were included.

Exclusion criteria were as follows: patients diagnosed with myofascial pain or muscle-related functional limitation; those who had previously undergone intra-articular injection or other invasive procedures involving the TMJ; patients with connective tissue diseases such as rheumatoid arthritis or with neurological disorders; patients with a history of major jaw trauma; and individuals with psychiatric disorders or a history of substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-12-13 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
The measurement of pain-free maximum mouth opening (MMO) in millimeters | Preopretive, Postoperative 1st day, 1st week and 1st month
  Pain-free MMO was measured as the distance between the incisal edges of the upper and lower incisors while patient's mouth is open as possible without any assistance and without pain. Three measurements were performed, and their average is recorded.
Change in post-operative pain assessed | Preoperative, Postoperative 1st day, 1st week and 1st month
  A visual analog scale (VAS) was used, grading from 1 to 10 (1: no pain, 10: unbearable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Eskişehir Osmangazi University, Eskişehir, Turkey (Türkiye)

REFERENCES:
- [Background] Hasanoglu Erbasar GN, Senturk MF, Sancak K. The Short-Term Results of the Modified Concentric-Needle Technique for Single-Puncture Arthrocentesis: A Preliminary Study. J Coll Physicians Surg Pak. 2024 Jun;34(6):717-722. doi: 10.29271/jcpsp.2024.06.717. PMID 38840358
- [Background] Senturk MF, Yazici T, Gulsen U. Techniques and modifications for TMJ arthrocentesis: A literature review. Cranio. 2018 Sep;36(5):332-340. doi: 10.1080/08869634.2017.1340226. Epub 2017 Jun 15. PMID 28618972